CLINICAL TRIAL: NCT06922929
Title: A Multicenter, Open-label, Prospective Phase III Clinical Trial to Evaluate the Diagnostic Efficacy and Safety of INR101 Injection for PET/CT Imaging in Participants With Suspected Recurrent Prostate Cancer After Radical Treatment
Brief Title: A Multicenter, Open-label, Prospective Phase III Clinical Trial to Evaluate INR101 Injection for PET/CT Imaging in Participants With Suspected Recurrent Prostate Cancer After Radical Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yunhe Pharmaceutical (Tianjin) Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INR101-III-01; CTR20250776 (Other: CDE)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer Recurrent
Keywords: suspected recurrent prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INR101 PET/ CT (Experimental): Drug: INR101 7±15% mCi of INR101 will be injected intravenously prior to perform the PET/CT
  Interventions: Drug: INR101

INTERVENTIONS:
Drug: INR101 — INR101 PET/ CT

SUMMARY:
A multicenter, open-label, prospective Phase III clinical trial to evaluate INR101 injection for PET/CT imaging in participants with suspected recurrent prostate cancer after radical treatment.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single-arm, non-randomized Phase III clinical trial evaluating the diagnostic efficacy and safety of INR101 injection PET/CT imaging in participants with suspected recurrence prostate cancer, who have experienced an increase in PSA levels after previously receiving radical treatment.

Participants enrolled in clinical trial will receive a single intravenous injection of INR101 injection at a dose of 7 mCi ± 15%, and PET/CT imaging will be performed 80 to 120 minutes after the injection.

The PET/CT images of INR101 injection for each participant will be interpreted independently by two readers blinded to all participant information. When the conclusions of the two readers are inconsistent, a third reader will be added for an adjudication interpretation (the third reader will also be in a blinded during the interpretation process and shall not be aware of the conclusions of the first two readers).

This study adopts a composite diagnostic criterion as the standard of truth. The interpretation of the composite diagnostic criterion is as follows: If a pathological diagnosis can be obtained, the pathological diagnosis shall be regarded as the standard of truth; if a pathological diagnosis cannot be obtained, a comprehensive interpretation shall be made based on the participant's medical history, changes in PSA levels and the results of conventional imaging examinations. The interpretation of the composite diagnostic criterion for each participant will be interpreted independently by two readers. When the conclusions of the two readers are inconsistent, a third reader will be added for an adjudication interpretation.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥18 years old
2. ECOG score of 0 or 1
3. Participants confirmed as prostate adenocarcinoma by histological pathological diagnosis, and have an elevated PSA level and are suspected of recurrence after previously receiving radical prostatectomy and/or radical radiotherapy (the PSA level is ≥ 0.2 ng/mL in two consecutive tests after 6 weeks following radical prostatectomy; or the PSA level is increased by ≥ 2 ng/mL compared to the lowest value after radical radiotherapy).
4. Routine blood tests, liver and kidney function meet the corresponding conditions:

   * Hemoglobin > 80 g/L; Platelet count > 50×10⁹/L
   * AST, ALT≤ 5 x ULN
   * Total bilirubin≤ 3 x ULN
5. Life expectancy of at least 6 months as assessed by investigator
6. Agree to use contraceptive measures from the date of signing the informed consent form to 3 months after medication administration, and avoid sperm donation
7. The participant/legal authorized representative understands the purpose and procedures of the trial and signs the informed consent form

Exclusion Criteria:

1. Participants who are unable to complete the imaging as required
2. Having had ≥ 2 types of malignant tumors within 5 years prior to the first administration, with the exception of fully treated non-metastatic thyroid cancer, basal cell carcinoma of the skin, superficial squamous cell carcinoma of the skin, and superficial bladder cancer.
3. Participants in other interventional clinical trials and within 5 half-lives of the investigational medicinal product or participants in other interventional clinical trials before signing the informed consent form; or participants in clinical trials of radioactive therapeutic drugs before signing the informed consent form and the time from the drug withdrawal to the signing date of the informed consent form is less than 3 months.
4. Have received intravenous iodine contrast agent within 24 hours prior to the administration of INR101, or have received any high-density oral contrast agent within 5 days (except for those who, as judged by the investigator, have no residual contrast agent in the intestines; oral water-soluble contrast agents are acceptable).
5. Participants with a history of salivary gland diseases or Paget's disease; participants with a history of fracture within the past year
6. Participants with hip joint prostheses
7. Known allergy to the active ingredients of INR101 or its components
8. Investigators judge that there are any medical diseases or other conditions that may affect safety, compliance or may affect the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
With the composite diagnostic criteria as the standard of truth, the positive predictive value (PPV) at the participant level by PET/CT imaging with INR101 injection of lesion detection | 3~12 months after administration
  The positive predictive value (PPV) of the participant level will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against imaging, clinical follow-up, and histopathology when available

SECONDARY OUTCOMES:
With pathological diagnosis as the standard of truth, Correct Detection Rate (CDR), Correct Localization Rate (CLR) at the participant level by PET/CT imaging with INR101 injection of lesion detection | 3~12 months after administration
  The Correct Detection Rate (CDR), Correct Localization Rate (CLR) of the participant level will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against imaging, clinical follow-up, and histopathology when available
With pathological diagnosis as the standard of truth, the positive predictive value (PPV) at the regional level (prostate, pelvic lymph nodes, extra-pelvic lymph nodes, visceral/soft tissues, bone) by PET/CT imaging with INR101 injection of lesion detect | 3~12 months after administration
  The positive predictive value (PPV) of the regional level (prostate, pelvic lymph nodes, extra-pelvic lymph nodes, visceral/soft tissues, bone) will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against imaging, clinical follow-up, and histopathology when available
In the group with negative baseline conventional imaging, the detection rate (DR), correct detection rate (CDR), and positive predictive value (PPV) at the participant level by PET/CT imaging with INR101 injection of lesion detection | 3~12 months after administration
  The detection rate (DR), correct detection rate (CDR), and positive predictive value (PPV) of the participant level will be determined of INR101 injection PET/CT imaging for detection of lesion, confirming against imaging, clinical follow-up, and histopathology when available
Among participants with different baseline PSA levels, the positive predictive value (PPV) at the participant level of PET/CT imaging with INR101 injection | 3~12 months after administration
  The positive predictive value (PPV) will be evaluated on a per- participant basis, stratified by PSA values: 0.2~0.5, 0.5~1.0, 1.0 ~2.0, 2.0~5.0, ≥5.0ng/mL
Assess the consistency of the diagnosis of PET/CT images intra- and inter-reader | 3~12 months after administration
  The intra- and inter-reader performance will be evaluated by adjudication rate and accept rate
Evaluate the safety and tolerability, including adverse events (AE)/serious adverse events (SAE), vital signs, physical examinations, laboratory tests and 12-lead electrocardiograms | 7 days after administration
  Adverse events will be determined through clinical assessment and categorized by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hongcheng Shi, Principal Investigator — Fudan University; Jianming Guo, Principal Investigator — Fudan University
Locations (32):
- China (32):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No